CLINICAL TRIAL: NCT05183022
Title: Do Total 30 Sphere Contact Lenses Provide a Comfortable Wearing Experience All Day?
Brief Title: Total30 Sphere Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008004
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Contact Lens Complication; Dry Eye
Keywords: Total30 Sphere Contact Lenses; Comfort; Dryness; Visual Analog Scale Scores
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This prospective, one-month, three-visit study will refit all participants into Total30 Sphere contact lenses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Total30 Sphere Contact Lenses (Experimental): All qualified participants will be refit into Total30 Sphere contact lenses.
  Interventions: Device: Total30 Sphere Contact Lenses

INTERVENTIONS:
Device: Total30 Sphere Contact Lenses — Participants will be refit into Total30 Sphere contact lenses and followed for 1 month.
  Other Names: Lehfilcon A

SUMMARY:
The purpose of this study is to map comfort over the full wear day in established, asymptomatic, soft CL wearers who are refit in Total30 Sphere CLs.

DETAILED DESCRIPTION:
Contact lens (CL) wearers frequently face eye discomfort symptoms, especially towards the end of the wear day. This burdensome discomfort can unfortunately cause patients to remove their CLs before their desired wear time. While comfortable wear times vary from patient to patient, Terry et al. has suggested that patients should be able to comfortably wear their CLs for at least 12 hours per day for at least 6 days per week. Nevertheless, the literature currently lacks sufficient data to comment fully on the full day wear experience, which for many patients may be 16 or more hours per day, especially if they have demanding careers. One CL that has the potential to allow for all day comfort is the Total30 Sphere CLs, which is a new water gradient, monthly CL aimed at delivering all day comfort and visual performance. Thus, the purpose of this study is to map comfort over the full wear day in established, asymptomatic, soft CL wearers who are refit in Total30 Sphere CLs. These data are not only important for judging the performance of Total30 Sphere CLs, but they will provide some of the first insights into the full day CL wearing experience over one month.

ELIGIBILITY:
Inclusion Criteria:

* Current contact lens wearers who have 20/20 visual acuity or better
* Minimally symptomatic as based upon Contact Lens Dry Eye Questionnaire scores (≤10)
* Astigmatism better than or equal to 0.50 D in each eye
* Must have regularly worn 2 week or monthly contact lenses within the past 6 months
* Must provide a glasses prescription that is is less than 3 years old
* Willing to start wearing their contact lenses between 6:00 AM and 8:00 AM and wear their contact lenses until 11:00 PM each day

Exclusion Criteria:

* Past or Current hard CL use
* Any known systemic health conditions that are thought to alter tear film physiology
* History of viral eye disease
* History of ocular surgery
* History of severe ocular trauma
* Active ocular infection or inflammation
* Currently using isotretinoin-derivatives
* Currently using ocular medications
* Currently using rewetting drops or artificial tear
* Pregnant or breast feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pucker, OD, MS, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Total30 Sphere Contact Lenses
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult, 18- to 45-year-old, contact lens wearers who had 20/20 visual acuity or better and who were minimally symptomatic contact lens wearers were recruited. This was a single arm study, so no baseline analyses were performed.
Arm/Group | Total30 Sphere Contact Lenses
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Total30 Participants | 26.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 31
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Ocular Comfort
Description: A visual analog scale (VAS) was used to compare end of day ocular comfort at 16 hours of contact lens wear over the 1 month study (0 to 100 scale with 100 being best).
Time Frame: 1 month
Population: Total30 Contact Lens Wearing Participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total30 Sphere Contact Lenses
Number analyzed (Participants) | 48
units on a scale
  Day 1: Comfort at Hour 16 | 36.66 (19.11)
  Day 2: Comfort at Hour 16 | 38.06 (14.71)
  Day 3: Comfort at hour 16 | 33.68 (22.49)
  Day 4: Comfort at hour 16 | 39.36 (13.95)
  Day 5: Comfort at hour 16 | 31.26 (24.73)
  2 weeks: Comfort at hour 16 | 33.84 (23.15)
  1 month: Comfort at hour 16 | 33.21 (22.39)
Statistical Analysis 1: Comparison: Total30 Sphere Contact Lenses; Test type: Superiority; p = 0.07, ANOVA

ADVERSE EVENTS:
Time Frame: Each participant was enrolled in this clinical trial for 1 month. The trial consisted of 3 in person visits (baseline, 1 week, and 1 month).
Description: Subjects were seen by an eye care professional three different times during the 1 month study. They were put through standard eye exam measures and contact lenses were thoroughly checked for comfort prior to distribution.
Arm/Group | Total30 Sphere Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT05183022/Prot_SAP_ICF_000.pdf